CLINICAL TRIAL: NCT04062604
Title: The Evaluation of the Lower Limb Function After Femur Fracture's Operation Treatment
Acronym: ELLFF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Marcin Bednarek, Principal Investigator, Jagiellonian University
Other Study IDs: ELLFF1
Record Dates: First submitted 2019-04-14; First posted 2019-08-20 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Surgical Treatment
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Femur fracture: Stabilization of femur fracture according to the AO fundation guidelines
  Interventions: Other: surgery
- Hip alloplasty: Endoprothesis
  Interventions: Other: surgery
- Knee alloplasty: Endoprothesis
  Interventions: Other: surgery
- Knee arthroscopy: Resection of the meniscus lesion or anterior cruciatus ligamentum reconstruction
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — surgical treatment of femur fracture, hip and knee alloplasty, knee arthroscopy

SUMMARY:
The goal of this study is the evaluation of lower limb function and the quaility of life of the patients after femur fracture operation treatment. LLTQ (Lower-Limb Tasks Questionnaire), LEFS (Lower Extremity Funcional Scale), LLFI-10 (Lower Limb Functional Index - 10) and LLFI (Lower Limb Functional Index) will be used for all the patients.

DETAILED DESCRIPTION:
All four questionnaires (LLTQ, LEFS LLFI-10 and LLFI) will be translated and adopted to the Polish conditions. The detailed medical/ epidemiological history will be collected in each patient. The fracture will be assessed based on the x-ray examination and will be qualified according to AO classification. NRS (Numerical Rating Scale) will be used to assess the pain intensity. SF36, QoL, CSQ, COPE and HADS questionnaire will be used to evaluate patient's the quality of life (subjective assessment). First assessment will be done before operation and then after 3, 6, 12, 24 month postoperation treatment.

With this main study, there is a plan to assess not only femur fractures patients, but the investigators would like to have addtional groups of the patients with hip and knee allopasty and knee arthroscopy with slightly different follow-up period: before the oparation, 1 and 12 month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed Patient Informed Consent
* Patients planned for the surgical treatment

Exclusion Criteria: n.a.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients planned for the surgical interventions
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Subjective assessment of the lower limb function | 12 month
  Questionnaire, score scale - according to the description in questionnaire, lower score- worse outcome
Objective assessment of the lower limb function | 12 month
  Physical exam

SECONDARY OUTCOMES:
Subjective assessment of the lower limb function | 3, 6, 24 months
  Questionnaire, score scale - according to the description in questionnaire, lower score- worse outcome
Objective assessment of the lower limb function | 3, 6, 24 months
  Physical exam

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Bednarek, Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided